CLINICAL TRIAL: NCT06959862
Title: ACURATE Enhance Post Market Study
Status: Withdrawn | Type: Observational
Why Stopped: Boston Scientific made the decision to discontinue worldwide commercialization of the ACURATE valve platform.
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: S2532
Record Dates: First submitted 2025-04-28; First posted 2025-05-07 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Aortic Valve Stenosis; Aortic Valve Calcification; Aortic Diseases
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Valve, Calcification of; Aortic Diseases | interventions — Transcatheter Aortic Valve Replacement; Replantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Transcatheter Aortic Valve Implantation/Replacement — The device is placed in patients heart at the level of aortic valve through a transfemoral access from femoral groin as indicated in device IFU

SUMMARY:
The objective of the ACURATE Enhance study is to assess valve frame expansion and hemodynamics in a routine clinical setting when optimized procedural steps for valve implantation are followed.

DETAILED DESCRIPTION:
ACURATE Enhance is a prospective, open-label, single-arm, multicenter, post-market study in patients implanted with the ACURATE neo2™ Aortic Valve System (or future commercially available iteration) for the treatment of severe calcific aortic stenosis in a routine clinical setting.

A subject who provides an Informed Consent Form (ICF) approved by the Independent Ethics Committee (IEC) and signed by the subject or the subject's legally authorized representative is considered enrolled once an attempt is made to insert the ACURATE neo2 Delivery System. Up to 150 subjects will be enrolled.

Follow-up will occur at pre-discharge, 30 days, 6 months and 1 year post index procedure per standard of care. Visits are in-person at 30 days and 1 year. The 6 month visits is in-person (preferred) or via telephone interview.

ELIGIBILITY:
Inclusion Criteria:

* Subject has documented severe aortic stenosis and an aortic annulus size compatible with the ACURATE neo2 valve per the commercial IFU based on the center's assessment of pre-procedure diagnostic imaging, and is deemed suitable for treatment with the ACURATE neo2™ Aortic Valve System (or future commercially available iteration) as confirmed by the Case Review Committee [CRC].
* Subject (or legal representative) understands the study requirements and provides written informed consent (eg, IEC-approved ICF).
* Subject, family member, and/or legal representative agree(s) and subject is capable of returning to the study hospital for all study required follow-up visits.

Exclusion Criteria:

* Subject has a previously implanted bioprosthesis in the aortic position.
* Subject has a unicuspid or bicuspid aortic valve.
* Subject has either of the following:

  * Severe vascular disease that would preclude safe access (e.g., aneurysm with thrombus that cannot be crossed safely; marked tortuosity; significant narrowing of the abdominal aorta; severe unfolding of the thoracic aorta; or thick, protruding, ulcerated atheroma in the aortic arch), OR
  * Severe/eccentric calcification of the aortic annulus that would prevent safe implantation of the TAVI prosthesis.
* Subject has known hypersensitivity to contrast agents that cannot be adequately pre-medicated or to the individual components of the study valve (nickel, titanium, processed porcine pericardium, polyethylene terephthalate [PET]).
* Subject has eGFR <30 mL/min (chronic kidney disease stage IV or stage V).
* Subject is unwilling or unable to undergo study required follow-up visits.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with symptomatic heart disease due to severe native calcific aortic stenosis
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint: | Index procedure
  Proportion of patients who achieve target valve frame expansion* at the end of the index procedure when following optimized procedural steps.
  * "Target valve frame expansion" is defined as visual evidence of parallel commissure posts, as confirmed by an independent core laboratory evaluation of procedural angiogram.

SECONDARY OUTCOMES:
Secondary Endpoint | 30 days
  All-cause mortality (cardiovascular and non-cardiovascular), Stroke (disabling and non-disabling) and Rehospitalization* at 30 days.
  * Rehospitalization refers to procedure-related or valve-related hospitalization, and includes the following as defined by VARC-3: hospitalization for new complications, bioprosthetic valve dysfunction (such as valve thrombosis, endocarditis, structural valve deterioration, or non-structural valve dysfunction), or heart-failure related hospitalizations.

OTHER OUTCOMES:
Safety endpoints adjudicated by an independent Clinical Events Committee | Peri- and post-procedure, pre-discharge or 7 days (whichever comes first), and 30 days, 6 months, and 1 year
  * All-cause mortality (cardiovascular and non-cardiovascular)
  * Stroke (NeuroARC Type 1a-d; disabling and non-disabling stroke)
  * Myocardial infarction (periprocedural [≤48 hours post index procedure] and spontaneous [>48 hours post index procedure])
  * Hospitalization for procedure- or valve-related causes, including hospitalization for new complications, bioprosthetic valve dysfunction (such as valve thrombosis, endocarditis, structural valve deterioration, or non-structural valve dysfunction), or heart-failure related hospitalizations
  * Acute kidney injury (≤7 days post index procedure) Stage 3 or 4 (requiring temporary or permanent renal replacement therapy)
  * Bleeding (Type 2 [major] and Type 3 or 4 [life-threatening or disabling])
  * Vascular complications (major)
  * Access-related non-vascular complications (major)
  * Cardiac structural complications (major)
Additional safety endpoints adjudicated by an independent Clinical Events Committee | Peri- and post-procedure, pre-discharge or 7 days (whichever comes first), and 30 days, 6 months, and 1 year
  * Valve-related complications, including conversion to open surgery, unplanned use of mechanical circulatory support, and implantation of >1 transcatheter valve during index hospitalization
  * Valve malposition, including valve migration, valve embolization, or ectopic valve deployment
  * Transcatheter aortic valve (TAV)-in-TAV deployment
  * New permanent pacemaker implantation resulting from new or worsened conduction disturbances
  * New onset of atrial fibrillation or atrial flutter
  * Coronary obstruction (≤3 days post index procedure)
  * Ventricular septal perforation (≤3 days post index procedure)
  * Annular rupture (≤3 days post index procedure)
  * Cardiac tamponade (≤3 days post index procedure)
  * Prosthetic aortic valve thrombosis (clinically significant)
  * Prosthetic aortic valve endocarditis
Safety endpoints per VARC-3 | Post-procedure, 30 days and 1 year
  * VARC-3 Device Success (post-procedure)
  * VARC-3 Early Safety composite at 30 days
  * VARC-3 Clinical Efficacy at 1 year
New York Heart Association (NYHA) functional classification | baseline, pre-discharge/7 days, 30 days, and 1 year
  Classification of heart failure symptoms as evaluated by NYHA classification
Prosthetic Aortic Valve Performance as measured by transthoracic echocardiography (TTE) | Pre-discharge/7days, 30 days, and 1 year
  Effective orifice area (EOA), Mean and Peak aortic gradients, peak aortic velocity, and grade of aortic regurgitation/paravalvular leak (PVL).
Patient reported outcomes and health status | baseline, 30 days and 1-year
  Patient reported outcomes and health status as evaluated by the Kansas City Cardiomyopathy Quality of Life questionnairec (KCCQ) at baseline and at 30-day and 1-year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Rück, Principal Investigator — Karolinska Universitetssjukhuset, Enheten för kardiologi

IPD SHARING:
Plan to Share IPD: Undecided
The data and study protocol for this clinical trial may be made available to other researchers in accordance with the Boston Scientific Data Sharing Policy. (http://www.bostonscientific.com/en-US/data-sharing-requests.html)